CLINICAL TRIAL: NCT02919475
Title: A Multicenter, Randomized, Double-blind, PlacebO-controlled, Parallel-group Study to EValuate the Efficacy and Safety of JTE-051 Administered for 12 Weeks to Subjects With Active Rheumatoid Arthritis (MOVE-RA)
Brief Title: Study to Evaluate Efficacy, Safety and Tolerability of JTE-051 in Subjects With Active Rheumatoid Arthritis
Acronym: MOVE-RA
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Akros Pharma Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: AE051-G-13-003
Record Dates: First submitted 2016-09-27; First posted 2016-09-29 (Estimated); Results first posted 2021-06-14 (Actual); Last update posted 2021-06-14 (Actual); Status verified 2021-06

CONDITIONS: Rheumatoid Arthritis
Keywords: JTE-051; Active Rheumatoid Arthritis; Efficacy; Safety; Tolerability; Rheumatoid Arthritis
MeSH Terms: conditions — Arthritis, Rheumatoid

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes

ARMS (5):
- JTE-051 Dose 1 (Experimental): One dose of study drug by mouth daily for 12 weeks
  Interventions: Drug: JTE-051
- JTE-051 Dose 2 (Experimental): One dose of study drug by mouth daily for 12 weeks
  Interventions: Drug: JTE-051
- JTE-051 Dose 3 (Experimental): One dose of study drug by mouth daily for 12 weeks
  Interventions: Drug: JTE-051
- JTE-051 Dose 4 (Experimental): One dose of study drug by mouth daily for 12 weeks
  Interventions: Drug: JTE-051
- Placebo (Experimental): One dose of study drug by mouth daily for 12 weeks
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: JTE-051 — Active drug tablets containing JTE-051
  Arms: JTE-051 Dose 1; JTE-051 Dose 2; JTE-051 Dose 3; JTE-051 Dose 4
Drug: Placebo — Placebo tablets identical in appearance to the active drug tablets
  Arms: Placebo

SUMMARY:
This study will evaluate the efficacy, safety, tolerability and pharmacokinetics (PK) of JTE-051 administered for 12 weeks in subjects with active rheumatoid arthritis who are receiving background non-biologic disease-modifying anti-rheumatic drug therapy.

ELIGIBILITY:
Inclusion Criteria:

* A diagnosis of RA prior to the Screening Visit.
* Active disease despite ongoing therapy with up to two non-biologic disease-modifying anti-rheumatic drugs, including methotrexate at both the Screening and Baseline Visits.
* Screening hs-CRP ≥1.2 x upper limit of normal (ULN).

Exclusion Criteria:

* Prior/current exposure to biologic and/or kinase inhibitor therapy.
* Known history or presence of polyneuropathy of any cause and no presence of clinically active compression neuropathy, radiculopathy or plexopathy at the Screening Visit.
* Positive test results for human immunodeficiency (HIV) virus, hepatitis B virus or hepatitis C (HCV) virus at the Screening Visit.
* Positive drug of abuse and alcohol test results.
* History of a clinically-significant infection that required oral antimicrobial or antiviral therapy within 8 weeks prior to Day 1.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 260 (Actual)
Dates: Start 2016-09-14 (Actual); Primary Completion 2018-06-25 (Actual); Study Completion 2018-06-25 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Yoshiro Masuda, Study Chair — Akros Pharma Inc.
Locations (39):
- United States (4):
  - Tucson, Arizona
  - Upland, California
  - Clearwater, Florida
  - Hendersonville, Tennessee
- Argentina (6):
  - La Plata, Buenos Aires
  - San Fernando, Buenos Aires
  - Barrio Norte, Córdoba Province
  - San Miguel de Tucumán, Tucumán Province
  - Córdoba
  - San Juan
- Bulgaria (4):
  - Lom
  - Plovdiv
  - Sevlievo
  - Sofia
- Colombia (3):
  - Medellín, Antioquia
  - Bogotá, Cundinamarca
  - Cali, Valle del Cauca Department
- Mexico (5):
  - Mexicali, B.C.
  - Guadalajara, Jalisco
  - Mexico City, Mexico City
  - San Luis Potosí City, San Luis Potosí
  - Mérida, Yucatán
- Lima, Peru
- Poland (3):
  - Warsaw, Masovian Voivodeship
  - Bialystok, Podlaskie Voivodeship
  - Elblag
- Romania (3):
  - Bucharest
  - Iași
  - Târgu Mureş
- Russia (3):
  - Kazan'
  - Moscow
  - Saint Petersburg
- Ukraine (7):
  - Kharkiv
  - Kherson
  - Kyiv
  - Lviv
  - Sumy
  - Vinnytsia
  - Zaporizhzhia

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Written informed consent was obtained prior to performing any study-related procedures. A copy of the informed consent was provided to each subject enrolled in this study. To qualify for the study, subjects were required to satisfy defined criteria.
Pre-assignment Details: Following informed consent signing, screening procedures to confirm eligibility were performed.
  1. Total screened - 528 subjects
  2. Screen failure - 268 subjects
  3. Randomized Population - 259 subjects (excluded 1 randomized subject due to site scientific misconduct)
  4. Intent-to-Treat Population - 257 subjects (excluded 2 randomized subjects: 1 was not dosed and 1 had no post-dose measurement)
  5. Safety Population - 258 subjects (excluded 1 randomized subject: 1 was not dosed)
Groups:
- JTE-051 50 mg: JTE-051 50 mg orally once daily for 12 weeks
- JTE-051 100 mg: JTE-051 100 mg orally once daily for 12 weeks
- JTE-051 150 mg: JTE-051 150 mg orally once daily for 12 weeks
- JTE-051 200 mg: JTE-051 200 mg orally once daily for 12 weeks
- Placebo: Placebo orally once daily for 12 weeks
Period: Overall Study
Arm/Group | JTE-051 50 mg | JTE-051 100 mg | JTE-051 150 mg | JTE-051 200 mg | Placebo
Started | 52 | 52 | 52 | 51 | 52
Started Dosing | 51 | 52 | 52 | 51 | 52
Completed | 46 | 44 | 47 | 38 | 48
Not Completed | 6 | 8 | 5 | 13 | 4
Not completed — Adverse Event | 3 | 3 | 3 | 9 | 2
Not completed — Death | 0 | 1 | 0 | 0 | 0
Not completed — Lost to Follow-up | 0 | 0 | 0 | 1 | 0
Not completed — Withdrawal by Subject | 2 | 3 | 1 | 2 | 2
Not completed — Inclusion/Exclusion Criteria Not Met | 1 | 1 | 1 | 1 | 0

BASELINE CHARACTERISTICS:
Population: Baseline characteristics results are reported for the Intent-to-Treat (ITT) population: 257 subjects who received at least one dose of JTE-051 or placebo and had at least one post-baseline efficacy assessment during the double-blind treatment period.
Groups:
- Total: Total of all reporting groups
Arm/Group | JTE-051 50 mg | JTE-051 100 mg | JTE-051 150 mg | JTE-051 200 mg | Placebo | Total
Number analyzed (Participants) | 51 | 51 | 52 | 51 | 52 | 257
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0 | 0 | 0 | 0
  Between 18 and 65 years | 42 | 48 | 46 | 43 | 44 | 223
  >=65 years | 9 | 3 | 6 | 8 | 8 | 34
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 41 | 40 | 44 | 43 | 43 | 211
  Male | 10 | 11 | 8 | 8 | 9 | 46
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 27 | 27 | 26 | 27 | 26 | 133
  Not Hispanic or Latino | 24 | 24 | 26 | 24 | 26 | 124
  Unknown or Not Reported | 0 | 0 | 0 | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 8 | 8 | 6 | 7 | 3 | 32
  Asian | 0 | 0 | 0 | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0 | 0 | 0
  Black or African American | 0 | 0 | 0 | 0 | 0 | 0
  White | 31 | 34 | 31 | 34 | 33 | 163
  More than one race | 12 | 9 | 15 | 10 | 16 | 62
  Unknown or Not Reported | 0 | 0 | 0 | 0 | 0 | 0

OUTCOME MEASURES:

1. Primary Outcome: Percentage of Subjects Achieving at Least 20% Improvement From Baseline in American College of Rheumatology (ACR) Core Set Measures (ACR20 Response Rate) Compared to Placebo at End-of-treatment (EOT)
Description: Percentage of subjects achieving at least 20% improvement from baseline (ACR20) in tender and swollen joint counts (ACR core set measures 1 and 2) and at least 20% improvement from baseline in the 3 of the 5 remaining ACR core set measures at EOT (up to Week 12) compared to placebo.
  The ACR core set measures are:
  1. Tender joint count
  2. Swollen joint count
  3. Subject Assessment of arthritis pain
  4. Subject's Global Assessment of disease activity (SGA)
  5. Physician's Global Assessment of disease activity (PGA)
  6. Health Assessment Questionnaire Disability Index (HAQ-DI)
  7. Acute Phase Reactant (i.e., hs-CRP - high sensitivity C-reactive protein)
Time Frame: Up to 12 Weeks
Population: Subjects in the Intent-to-Treat (ITT) population (subjects who received at least one dose of JTE-051 or placebo, and had at least one post-baseline efficacy assessment during the double-blind treatment period) with available efficacy assessment(s) results at EOT (up to Week 12).
Measure: Count of Participants; unit: Participants
Arm/Group | JTE-051 50 mg | JTE-051 100 mg | JTE-051 150 mg | JTE-051 200 mg | Placebo
Number analyzed (Participants) | 51 | 51 | 50 | 51 | 52
Participants | 27 | 31 | 27 | 30 | 29
Statistical Analysis 1: Comparison: JTE-051 50 mg vs Placebo; Test type: Superiority; p = 0.842, Fisher Exact
Statistical Analysis 2: Comparison: JTE-051 100 mg vs Placebo; Test type: Superiority; p = 0.841, Fisher Exact
Statistical Analysis 3: Comparison: JTE-051 150 mg vs Placebo; Test type: Superiority; p = 0.842, Fisher Exact
Statistical Analysis 4: Comparison: JTE-051 200 mg vs Placebo; Test type: Superiority; p > 0.999, Fisher Exact

2. Secondary Outcome: Percentage of Subjects Achieving ACR20 Response Rate Compared to Placebo at Week 12
Description: Percentage of subjects achieving at least 20% improvement from baseline (ACR20) in tender and swollen joint counts (ACR core set measures 1 and 2) and at least 20% improvement from baseline in the 3 of the 5 remaining ACR core set measures at Week 12 compared to placebo.
  The ACR core set measures are:
  1. Tender joint count
  2. Swollen joint count
  3. Subject Assessment of arthritis pain
  4. Subject's Global Assessment of disease activity (SGA)
  5. Physician's Global Assessment of disease activity (PGA)
  6. Health Assessment Questionnaire Disability Index (HAQ-DI)
  7. Acute Phase Reactant (i.e., hs-CRP - high sensitivity C-reactive protein)
Time Frame: Week 12
Population: Subjects in the ITT population (subjects who received at least one dose of JTE-051 or placebo, and had at least one post-baseline efficacy assessment during the double-blind treatment period) with available efficacy assessment(s) results at Week 12.
Measure: Count of Participants; unit: Participants
Arm/Group | JTE-051 50 mg | JTE-051 100 mg | JTE-051 150 mg | JTE-051 200 mg | Placebo
Number analyzed (Participants) | 46 | 45 | 47 | 38 | 48
Participants | 26 | 28 | 25 | 24 | 28
Statistical Analysis 1: Comparison: JTE-051 50 mg vs Placebo; Test type: Superiority; p > 0.999, Fisher Exact
Statistical Analysis 2: Comparison: JTE-051 100 mg vs Placebo; Test type: Superiority; p = 0.832, Fisher Exact
Statistical Analysis 3: Comparison: JTE-051 150 mg vs Placebo; Test type: Superiority; p = 0.682, Fisher Exact
Statistical Analysis 4: Comparison: JTE-051 200 mg vs Placebo; Test type: Superiority; p = 0.665, Fisher Exact

3. Secondary Outcome: Percentage of Subjects Achieving ACR50 Response Rate Compared to Placebo at Week 12
Description: Percentage of subjects achieving at least 50% improvement from baseline (ACR50) in tender and swollen joint counts (ACR core set measures 1 and 2) and at least 50% improvement from baseline in the 3 of the 5 remaining ACR core set measures at Week 12 compared to placebo.
  The ACR core set measures are:
  1. Tender joint count
  2. Swollen joint count
  3. Subject Assessment of arthritis pain
  4. Subject's Global Assessment of disease activity (SGA)
  5. Physician's Global Assessment of disease activity (PGA)
  6. Health Assessment Questionnaire Disability Index (HAQ-DI)
  7. Acute Phase Reactant (i.e., hs-CRP - high sensitivity C-reactive protein)
Time Frame: Week 12
Population: as for outcome 2
Measure: Count of Participants; unit: Participants
Arm/Group | JTE-051 50 mg | JTE-051 100 mg | JTE-051 150 mg | JTE-051 200 mg | Placebo
Number analyzed (Participants) | 46 | 45 | 47 | 38 | 48
Participants | 10 | 12 | 8 | 11 | 10
Statistical Analysis 1: Comparison: JTE-051 50 mg vs Placebo; Test type: Superiority; p > 0.999, Fisher Exact
Statistical Analysis 2: Comparison: JTE-051 100 mg vs Placebo; Test type: Superiority; p = 0.627, Fisher Exact
Statistical Analysis 3: Comparison: JTE-051 150 mg vs Placebo; Test type: Superiority; p = 0.794, Fisher Exact
Statistical Analysis 4: Comparison: JTE-051 200 mg vs Placebo; Test type: Superiority; p = 0.453, Fisher Exact

4. Secondary Outcome: Percentage of Subjects Achieving ACR70 Response Rate Compared to Placebo at Week 12
Description: Percentage of subjects achieving at least 70% improvement from baseline (ACR70) in tender and swollen joint counts (ACR core set measures 1 and 2) and at least 70% improvement from baseline in the 3 of the 5 remaining ACR core set measures at Week 12 compared to placebo.
  The ACR core set measures are:
  1. Tender joint count
  2. Swollen joint count
  3. Subject Assessment of arthritis pain
  4. Subject's Global Assessment of disease activity (SGA)
  5. Physician's Global Assessment of disease activity (PGA)
  6. Health Assessment Questionnaire Disability Index (HAQ-DI)
  7. Acute Phase Reactant (i.e., hs-CRP - high sensitivity C-reactive protein)
Time Frame: Week 12
Population: as for outcome 2
Measure: Count of Participants; unit: Participants
Arm/Group | JTE-051 50 mg | JTE-051 100 mg | JTE-051 150 mg | JTE-051 200 mg | Placebo
Number analyzed (Participants) | 46 | 45 | 47 | 38 | 48
Participants | 3 | 5 | 4 | 4 | 0
Statistical Analysis 1: Comparison: JTE-051 50 mg vs Placebo; Test type: Superiority; p = 0.113, Fisher Exact
Statistical Analysis 2: Comparison: JTE-051 100 mg vs Placebo; Test type: Superiority; p = 0.024, Fisher Exact
Statistical Analysis 3: Comparison: JTE-051 150 mg vs Placebo; Test type: Superiority; p = 0.056, Fisher Exact
Statistical Analysis 4: Comparison: JTE-051 200 mg vs Placebo; Test type: Superiority; p = 0.035, Fisher Exact

5. Secondary Outcome: Change From Baseline in SDAI (Simplified Disease Activity Index) at Week 12
Description: The SDAI Scores indicate how active a patient's rheumatoid arthritis (RA) is currently. The SDAI is the sum of 5 outcome parameters: tender joint score (0 to 28), swollen joint score (0 to 28), Patient's Global Score of disease activity (0 to 10), Physician's Global Score of disease activity (0 to 10) and C-reactive protein (CRP, 0 to 10).General SDAI Score Interpretation is as follows:
  0.0 - 3.3 Remission 3.4 - 11.0 Low Activity 11.1 - 26.0 Moderate Activity 26.1 - 86.0 High Activity
Time Frame: Week 12
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: Score on a scale
Arm/Group | JTE-051 50 mg | JTE-051 100 mg | JTE-051 150 mg | JTE-051 200 mg | Placebo
Number analyzed (Participants) | 46 | 45 | 46 | 38 | 48
Score on a scale | -18.14 (15.437) | -21.68 (13.275) | -19.41 (16.446) | -19.97 (14.244) | -17.66 (16.816)

6. Secondary Outcome: Change From Baseline in CDAI (Clinical Disease Activity Index) at Week 12
Description: The CDAI is a useful clinical composite score for following patients with rheumatoid arthritis (RA). The CDAI is the sum of 4 outcome parameters: tender joint score (0 to 28), swollen joint score (0 to 28), Patient's Global Score of disease activity (0 to 10) and Physician's Global Score of disease activity (0 to 10). The CDAI Score Interpretation is as follows:
  0 to 2.8: Remission 2.9 to 10: Low Disease Activity 10.1 to 22: Moderate Disease Activity 22.1 to 76: High Disease Activity
Time Frame: Week 12
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: Score on a scale
Arm/Group | JTE-051 50 mg | JTE-051 100 mg | JTE-051 150 mg | JTE-051 200 mg | Placebo
Number analyzed (Participants) | 46 | 45 | 47 | 38 | 48
Score on a scale | -18.76 (14.768) | -22.40 (13.469) | -21.02 (16.153) | -21.24 (14.208) | -17.19 (15.548)

7. Secondary Outcome: Change From Baseline in DAS28-CRP (Disease Activity Score [DAS] Based on High-sensitivity C-reactive Protein [Hs-CRP]) at Week 12
Description: Disease Activity Score (DAS) modified to include 28 joint count (DAS28) consists of composite score of following variables: 28 tender joint count (TJC28) ranging from 0 to 28, 28 swollen joint count (SJC28) ranged from 0 to 28, C-reactive protein (CRP) (milligrams per liter) and subject's global assessment of disease activity (SGA) ranging from 0 (no disease activity) to 10 (extremely active disease). DAS28-CRP was calculated using following formula:
  DAS28-CRP=0.56*square root (sqrt)(TJC28)+0.28*sqrt(SJC28)+0.36*natural log(CRP+1)+0.014*SGA+0.96.
  DAS28-CRP ranged from 0.96-9.4, where lower scores indicated less disease activity and remission is DAS28-CRP <2.6.
  A decrease in DAS28-CRP indicated an improvement in participant's condition.
Time Frame: Week 12
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: Score on a scale
Arm/Group | JTE-051 50 mg | JTE-051 100 mg | JTE-051 150 mg | JTE-051 200 mg | Placebo
Number analyzed (Participants) | 46 | 45 | 46 | 38 | 48
Score on a scale | -0.95 (1.039) | -1.23 (0.979) | -1.03 (1.123) | -1.10 (0.987) | -0.98 (1.123)

8. Secondary Outcome: Change From Baseline in HAQ-DI (Health Assessment Questionnaire Disability Index) at Week 12
Description: The HAQ-DI questionnaire assesses the participant's self-perception on the degree of difficulty [0 (without any difficulty), 1 (with some difficulty), 2 (with much difficulty), and 3 (unable to do)] in 8 functional area categories: (1) dressing and grooming; (2) arising; (3) eating; (4) walking; (5) hygiene; (6) reaching; (7) gripping; and (8) performing other daily activities. Scores from each functional area category (total 8 categories) were averaged to calculate the HAQ-DI score, which ranged from 0 (no disability) to 3 (severe disability). A decrease in HAQ-DI score indicated an improvement in the participant's condition.
Time Frame: Week 12
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: Score on a scale
Arm/Group | JTE-051 50 mg | JTE-051 100 mg | JTE-051 150 mg | JTE-051 200 mg | Placebo
Number analyzed (Participants) | 46 | 45 | 47 | 38 | 48
Score on a scale | -0.52 (0.600) | -0.71 (0.629) | -0.60 (0.620) | -0.80 (0.727) | -0.47 (0.616)

9. Secondary Outcome: Number of Subjects With Treatment-related Adverse Events
Description: Subjects in the Safety Population (258, subjects who were randomly assigned to treatment and who received at least one dose of study drug). The number of subjects in the Safety Population is 258 subjects, which is 1 less than the Randomized Population of 259 subjects, since 1 randomized subject did not receive any study drug.
Time Frame: Up to 16 Weeks
Population: Subjects in the Safety Population (258, subjects who were randomly assigned to treatment and who received at least one dose of study drug). The number of subjects in the Safety Population is 258 subjects, which is 1 less than the Randomized Population of 259 subjects, since 1 randomized subject did not receive any study drug.
Measure: Count of Participants; unit: Participants
Arm/Group | JTE-051 50 mg | JTE-051 100 mg | JTE-051 150 mg | JTE-051 200 mg | Placebo
Number analyzed (Participants) | 51 | 52 | 52 | 51 | 52
Participants
  Number of subjects with TEAEs | 26 | 21 | 32 | 34 | 22
  Number of subjects with no TEAEs | 25 | 31 | 20 | 17 | 30

10. Secondary Outcome: Trough Concentrations (Ctrough) of JTE-051 in Plasma at Week 12
Time Frame: Week 12
Population: Subjects in the Pharmacokinetic (PK) population (received at least one dose of JTE-051 and have at least one usable JTE-051 plasma concentration measurement) with available trough plasma concentrations of JTE-051 at Week 12.
Measure: Mean (Standard Deviation); unit: ng/mL
Arm/Group | JTE-051 50 mg | JTE-051 100 mg | JTE-051 150 mg | JTE-051 200 mg
Number analyzed (Participants) | 40 | 42 | 40 | 35
ng/mL | 119 (96.9) | 178 (156) | 312 (252) | 354 (281)

ADVERSE EVENTS:
Time Frame: Up to 16 weeks
Description: The Safety Population (258, subjects who were randomly assigned to treatment and who received at least one dose of study drug) was used for safety analysis. The number of subjects in the Safety Population is 258 subjects, which is 1 less than the Randomized Population of 259 subjects, since 1 randomized subject did not receive any study drug.
Arm/Group | JTE-051 50 mg | JTE-051 100 mg | JTE-051 150 mg | JTE-051 200 mg | Placebo
All-Cause Mortality (participants affected / at risk) | 0/51 | 1/52 | 0/52 | 0/51 | 0/52
Serious Adverse Events (participants affected / at risk) | 2/51 | 3/52 | 2/52 | 1/51 | 0/52
Other Adverse Events (participants affected / at risk) | 11/51 | 7/52 | 20/52 | 21/51 | 3/52
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | JTE-051 50 mg (N=51) | JTE-051 100 mg (N=52) | JTE-051 150 mg (N=52) | JTE-051 200 mg (N=51) | Placebo (N=52)
Abdominal pain/Diffused abdominal pain (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Gastric ulcer (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Appendicitis (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Cellulitis/Cellulitis in right hand (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Pneumonia/Bilateral pneumonia (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) — This serious adverse event resulted in death (assessed as not related).
Rheumatoid arthritis/Exacerbation of rheumatoid arthritis (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Insomnia/Sleep Disorders: Insomnia (Psychiatric disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Urticaria (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | JTE-051 50 mg (N=51) | JTE-051 100 mg (N=52) | JTE-051 150 mg (N=52) | JTE-051 200 mg (N=51) | Placebo (N=52)
Anemia (Blood and lymphatic system disorders) | 1 (1) | 1 (1) | 3 (3) | 2 (2) | 1 (1)
Constipation (Gastrointestinal disorders) | 3 (3) | 1 (1) | 6 (6) | 2 (2) | 0 (0)
Nasopharyngitis (Infections and infestations) | 2 (2) | 1 (1) | 4 (4) | 0 (0) | 0 (0)
Urinary tract infection (Infections and infestations) | 3 (3) | 3 (3) | 5 (5) | 8 (8) | 2 (2)
Dysgeusia (Nervous system disorders) | 2 (2) | 1 (1) | 2 (2) | 9 (9) | 0 (0)

LIMITATIONS AND CAVEATS:
None reported.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The sponsor can review results communications at least 60 days prior to public release. The sponsor will have a review period of 60 days and can embargo communications regarding trial results for an additional period of 60 days from the end of sponsor review period. The sponsor may require removal of any and all confidential information (other than study results) in the communication.

DOCUMENTS (2):
  • Study Protocol (2016-03-24): https://cdn.clinicaltrials.gov/large-docs/75/NCT02919475/Prot_000.pdf
  • Statistical Analysis Plan (2018-08-10): https://cdn.clinicaltrials.gov/large-docs/75/NCT02919475/SAP_001.pdf